CLINICAL TRIAL: NCT04068311
Title: Implementation of Multidisciplinary Assessments for Geriatric Patients in an Emergency Department Observation Unit
Brief Title: Implementation of Multidisciplinary Assessments for Geriatric Patients in an ED Observation Unit
Acronym: IMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lauren Southerland, Associate Professor, Department of Emergency Medicine, Ohio State University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2019H0109; K23AG061284-01A1 (NIH)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Fall Patients; Delirium; Quality of Life; Functional Status
Keywords: Geriatrics; Emergency Medicine; Implementation; Consolidated Framework for Implementation Research
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Pre and post cohort study with an intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre Implementation (No Intervention): Adult patients >65 years of age in the Emergency Department Observation Unit.
- Post Implementation (Active Comparator): Adult patients >65 years of age in the Emergency Department Observation Unit.
  Interventions: Other: Geriatric Screening tools

INTERVENTIONS:
Other: Geriatric Screening tools — Lean Six Sigma implementation in the Emergency Department of nurse-driven geriatric screening tools and protocols for patients with fall risk, delirium, and high risk scores.
  Arms: Post Implementation

SUMMARY:
This project will implement a 2 step protocol for multidisciplinary geriatric assessment in the Emergency Department (ED). Candidate: Dr. Lauren Southerland is a Geriatric- and Emergency Medicine-trained physician at The Ohio State University Wexner Medical Center. Training: The career development plan will build upon Dr. Southerland's unique fellowship training in Geriatrics with courses in Implementation and Dissemination Science, a Black Belt in Lean Six Sigma, and Master's in Public Health courses. This combination will position her as an expert in Implementation research, with the career goal of translating validated, effective elements of geriatric care into the daily practice of Emergency Medicine. Mentors: Dr. Southerland has an experienced mentorship team who will provide guidance in the intricacies of emergency research (Dr. Jeffrey Caterino, MD, MPH), implementation strategies and studies of hospital staff and nurses (Dr. Lorraine Mion, PhD), implementation frameworks and reporting (Dr. Christopher Carpenter, an emergency medicine physician at Washington University at St. Louis), and identifying environmental and human factor barriers to quality care. Project: Multidisciplinary assessment by geriatricians, physical therapists, case managers, and pharmacists identifies and addresses underlying geriatric issues in older ED patients. However, only a few EDs across the country have been able to incorporate multidisciplinary care for their older patients, due to barriers such as personnel costs, work flow culture, and the 24 hour ED care model. We developed a two-step protocol to address these barriers: Step 1 is quick, sensitive screens for fall risk (4 Stage Balance Test), delirium (Brief Delirium Triage Screen), and frailty (Identifying Seniors at Risk Score). Patients with concerning results will be placed in an ED Observation Unit for (step 2) multidisciplinary geriatric assessment. In Aim 1 we will use the Consolidated Framework for Implementation Research and Lean Six Sigma methods to identify and address residual barriers to full implementation. Aim 2 will evaluate the effectiveness of this protocol in regards to patient-oriented outcomes (functional status and health-related quality of life at 90 days). By using implementation frameworks and processes, we will develop a protocol that is effective, sustainable, and ready for dissemination to EDs across the US.

DETAILED DESCRIPTION:
Older adult patients in the Emergency Department frequently experience poor outcomes due to lack of recognition of underlying syndromes, such as delirium, polypharmacy, falls, and social needs. This study uses rigorous implementation science processes to implement and investigate an ED protocol to screen older adults for these syndromes and address them with multidisciplinary geriatric assessments in an ED Observation Unit. Using an Observation Unit to evaluate older adult patients at risk is a novel strategy developed to address the current barriers of sustainability, cost, and timeliness that arose in prior studies of geriatric assessments in an ED setting.

Specific Aim 1: Implementation: Develop, implement, and sustain a two-step intervention providing ED geriatric assessments by combining 1) ED nurse-based screening for geriatric syndromes of all older ED patients with 2) multidisciplinary geriatric assessment in an ED Obs Unit. Mixed-methods approaches and the Consolidated Framework for Implementation (CFIR) will be used to identify resource, organizational, patient, staff, and administrative factors that affect protocol adherence. Lean Six Sigma processes will be used to overcome barriers. The effects of the protocol in reference to ED quality metrics, staff work flow, and work culture will be tracked.

Hypothesis 1a: Implementation: Lean Six Sigma processes will i) increase ED nurse-based screening rates to >80% older adults in the ED and ii) increase protocol fidelity in the Obs Unit to >80%.

Hypothesis 1b: Sustainability: After 6 months of >80% screening, the investigators will characterize the necessary elements for sustainability by systematically withdrawing implementation support strategies. Hypothesis: Attention to CFIR elements during implementation will result in routinization and institutionalization that does not significantly decrease with withdrawal or time, as assessed by sustainability surveys.37

Specific Aim 2: Effectiveness: The investigators will describe the effect of this protocol on reducing the decline in functional status and reducing other patient and systems outcomes (e.g. health related quality of life (HRQoL)) commonly seen after an ED visit.38-40 To obtain patient-centered outcomes, two patient cohorts (pre and post implementation) will be recruited.

Hypothesis 2a: The intervention will reduce the decline in functional status seen after ED visits. Secondary outcomes include health-related quality of life, ED revisits, and results of the multidisciplinary assessments.

Hypothesis 2b: Patients will be satisfied with the protocol as assessed by thematic analysis of qualitative subject interviews of post intervention patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 65 years old assigned to the Emergency Department Observation Unit for care

Exclusion Criteria:

* need for inpatient care at the time of initial Emergency Department disposition
* non-English speaking
* acute psychiatric issues requiring stabilization by psychiatry team
* prisoners
* unable to consent and no legally authorized representative available.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 373 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Southerland, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Southerland LT, Stephens JA, Hunold KM, Carpenter CR, Mion LC, Krupinski L, Reider CR, Caterino JM. Effects of a Geriatric Emergency Department Multidisciplinary Intervention on Functional Status and Quality of Life: A Pre/Post Cohort Study. Acad Emerg Med. 2026 Jan;33(1):e70119. doi: 10.1111/acem.70119. Epub 2025 Aug 6. PMID 40770643
- [Derived] Southerland LT, Stephens JA, Carpenter CR, Mion LC, Moffatt-Bruce SD, Zachman A, Hill M, Caterino JM. Study protocol for IMAGE: implementing multidisciplinary assessments for geriatric patients in an emergency department observation unit, a hybrid effectiveness/implementation study using the Consolidated Framework for Implementation Research. Implement Sci Commun. 2020 Feb 25;1:28. doi: 10.1186/s43058-020-00015-7. eCollection 2020. PMID 32885187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the pre-implementation cohort occurred Sep 2019 - Nov 2020. Recruitment was terminated early due to external pressures [we were at risk of losing accreditation as a Level 1 Geriatric emergency department if we did not show progress]. Implementation roll out was paused until March 2021 due to the COVID-19 pandemic. The implementation period was March 2021-August 2022. The post-implementation cohort enrolled from Sep 2022-Aug 2023.
Groups:
- Pre-Implementation Cohort: Cohort of participants enrolled prior to the implementation of geriatric screening throughout the Emergency Department
- Post-Implementation Cohort: A cohort of participants enrolled after geriatric screening was implemented in the Emergency Department
Period: Overall Study
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Started | 143 (Goal recruitment 150) | 230 (Goal recruitment 230)
Recruited | 143 | 230
Analysis set | 138 | 230
Completed | 111 | 159
Not Completed | 32 | 71
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 24 | 68
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort | Total
Number analyzed (Participants) | 138 | 230 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (6.5) | 73.2 (6.4) | 73.3 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 120 | 187
  Male | 71 | 110 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 136 | 229 | 365
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 18 | 28 | 46
  White | 114 | 196 | 310
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 3 | 6
Charlson Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — The Charlson Comorbidity Index is a weighted scale using the previous diseases (comorbidities) that a patient has to give an estimate of their overall burden of illness. The score ranges from 0-37 points with 0 being no significant comorbidities and 37 being the highest comorbidity burden.
  units on a scale | 5.2 (2.65) | 4.79 (2.06) | 4.9 (2.3)
Global Physical Health Quality of Life score (PROMIS) [Mean (Standard Deviation); unit: T score] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2 is a 10-item patient-reported questionnaire assessing overall health and well-being. It provides two summary scores: Global Physical Health and Global Mental Health. Each of the two scores are standardized to the general US population, with a mean of 50 and a standard deviation of 10. Higher scores indicate better physical health. This measure is reported in raw scores of 4 to 20 (range), with T scores of 1 to 99. This section reports the Global Physical Health score.
  T score | 43.9 (8.4) | 45.1 (8.4) | 44.6 (8.4)
Global Mental Health Quality of Life score (PROMIS) [Mean (Standard Deviation); unit: T score] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2 is a 10-item patient-reported questionnaire assessing overall health and well-being. It provides two summary scores: Global Physical Health and Global Mental Health. Each of the two scores are standardized to the general US population, with a mean of 50 and a standard deviation of 10. Higher scores indicate better physical or mental health. This measure is reported in raw scores of 4 to 20 (range), with T scores of 1-99. This section reports the Global Mental Health score.
  T score | 49.6 (8.0) | 50.8 (8.1) | 50.4 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life (HRQoL) Using the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2 is a 10-item patient-reported questionnaire assessing overall health and well-being. It provides two summary scores: Global Physical Health and Global Mental Health. Each of the two scores are standardized to the general US population, with a mean of 50 and a standard deviation of 10. Higher scores indicate better physical or mental health. This measure is reported in raw scores of 4 to 20 (range), with T scores of 16.2 - 67.7.
Time Frame: 90 days
Population: Change in HRQoL at 90 days was obtained by subtracting the t-score from day 0 to day 90 for each participant and comparing both cohorts. Therefore we changed the t scores to a delta in scores and report mean and standard deviation of the change.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Number analyzed (Participants) | 111 | 161
T score | -0.73 (6.98) | -0.33 (5.46)
Statistical Analysis 1: Comparison: Pre-Implementation Cohort vs Post-Implementation Cohort; Test type: Superiority; p = 0.61, Chi-squared

2. Secondary Outcome: Functional Status Using OARS: Older Americans Resources and Services Program Activities of Daily Living, Independent Activities of Daily Living Summary Scale
Description: We report the number of participants with a decrease of 3 points or more, our definition of functional decline. The OARS: Older Americans Resources and Services Program Activities of Daily Living Score ranges from 0-28, with higher scores representing worsening functional status. A change of 3 points is considered clinically significant functional decline.
Time Frame: 90 days
Population: We defined a significant decline in Functional Status (OARS) as decrease of 3 or more points from day 0 to day 90. Comparisons between the pre and post cohorts were done using either Chi-square tests for proportions. A multivariable logistic regression model was planned to compare outcomes between the groups while controlling for any significant factors varying between the two cohorts, but was not able to be done due to the low number of primary outcome events.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Number analyzed (Participants) | 111 | 159
Participants | 4 | 5
Statistical Analysis 1: Comparison: Pre-Implementation Cohort vs Post-Implementation Cohort; Test type: Superiority; p = 0.83, Chi-squared — unadjusted

3. Secondary Outcome: Number of Participants Who Received Home Resources, Services and/or New Diagnoses of Geriatric Syndromes
Description: Numerical tally of the outcomes of multidisciplinary geriatric assessment- arrangement for new home resources such as medical equipment and mobility equipment, new services such as home health, and new diagnoses of geriatrics syndromes.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Number analyzed (Participants) | 138 | 230
Participants | 33 | 67
Statistical Analysis 1: Comparison: Pre-Implementation Cohort vs Post-Implementation Cohort; Test type: Superiority; p = 0.14, Chi-squared

4. Secondary Outcome: Geriatric Screening Rates
Description: Percentage of older adults in the Emergency Department who are screened for geriatric syndromes with the Identifying Seniors at Risk tool, the brief delirium triage screen, and the 4 Stage Balance Test
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
Number analyzed (Participants) | 138 | 230
Participants | 17 | 210
Statistical Analysis 1: Comparison: Pre-Implementation Cohort vs Post-Implementation Cohort; Test type: Superiority; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Pre-Implementation Cohort | Post-Implementation Cohort
All-Cause Mortality (participants affected / at risk) | 3/143 | 3/230
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/230
Other Adverse Events (participants affected / at risk) | 0/143 | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04068311/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT04068311/ICF_001.pdf